CLINICAL TRIAL: NCT00301106
Title: Phase I Trial of Adenoviral Vector Delivery of the Human Interleukin-12 cDNA by Intratumoral Injection in Patients With Metastatic Breast Cancer to the Liver
Brief Title: Biological Therapy in Treating Women With Breast Cancer That Has Spread to the Liver
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: protocol underwent significant revisions, decision made to terminate study and open as new study listed NCT00849459
Sponsor: Max Sung (Other)
Responsible Party: Sponsor-Investigator, Max Sung, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 97-779; MTS-GCO-97-779; MTS-9911-358; MTS-A-8200; CDR0000456626
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: stage IV breast cancer; liver metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenovirus-mediated human interleukin-12 (Experimental): starting dose of ADV-hIL12 - 1 x 10 to the 10th power vp (virus particles) per patient, escalating in half-log increments up to 1 x 10 to the 13th power vp per patient, after which dose escalation will be at lower increments of 2 x 10 to the 13th power vp, to a maximum of 3.0 x 10 to the 13th power vp per patient.
  Interventions: Biological: adenovirus-mediated human interleukin-12

INTERVENTIONS:
Biological: adenovirus-mediated human interleukin-12 — The purified ADV-hIL12 is suspended in formulation buffer (10mM Tris, pH 7.5/
  1mM MgCl2/ 150mM NaCl/ 10% glycerol) and aliquoted into 1ml cryovials. The filled vials are stored at or below -60 degC.

SUMMARY:
RATIONALE: Biological therapy using a gene-modified virus that can make interleukin-12 may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of a gene-modified virus that can make interleukin-12 in treating women with breast cancer that has spread to the liver.

DETAILED DESCRIPTION:
Direct intratumoral injection of metastatic hepatic tumors using an adenoviral vector expressing the human recombinant interleukin-12 gene (Adv.RSV-hIL12, also termed ADV-hIL-12).

OBJECTIVES:

* Study the toxicity of escalating doses of adenoviral vector expressing the human recombinant interleukin-12 gene, administered by percutaneous intratumoral injection, in women with liver metastasis secondary to breast cancer.
* Determine tumor responses produced by this regimen.
* Determine immune responses induced by this regimen.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed* breast adenocarcinoma metastatic to the liver

  * Solitary or multiple hepatic metastases

    * No malignant involvement of > 40% of the estimated liver volume NOTE: *Must be from the hepatic tumor designated for study injection
* Metastatic liver tumors must be measurable in ≥ 2 dimensions on CT scan or MRI
* At least 1 metastatic hepatic tumor ≥ 2 cm in diameter must be visualized by ultrasound and accessible for percutaneous injection under ultrasound guidance
* Extrahepatic metastasis allowed
* No solitary hepatic metastasis eligible for liver resection
* No clinical evidence for severe liver disease (e.g., prior or current ascites or portosystemic encephalopathy)
* Hormone-receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Granulocyte count ≥ 1,500/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm^3
* PT ≤ 14.5 sec
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 45 mL/min
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Transaminases ≤ 2.5 times ULN
* Karnofsky performance status ≥ 70%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after completion of study treatment
* No active infection or serious intercurrent medical illness
* No HIV infection
* Life expectancy ≥ 16 weeks
* No other malignancy within the past 5 years except inactive nonmelanoma skin cancer, in situ carcinoma of the cervix, or grade 1 papillary bladder cancer
* At highest dose level, patient must weigh ≥ 30 kg

PRIOR CONCURRENT THERAPY:

* No systemic immunosuppressive drugs, including corticosteroids, within 2 months prior to study entry

  * Not require immunosuppressive drugs or anticoagulant therapy with heparin or warfarin for at least 2 months after study treatment
* No chemotherapy within 4 weeks of study entry (6 weeks for nitrosoureas)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Toxicity | up to 15 days
  Serial monitoring of tumor necrosis factor alpha (TNFα) levels

SECONDARY OUTCOMES:
Tumor Response | up to 2 months
  Sequential assessment of tumor on CT or MRI
IL12 level Immune response | up to 2 months
  Serum IL12 level
IFNγ levels Immune response | up to 2 months
  IFNγ levels
Immune response | up to 2 months
  Serum antibodies (titer) to adenovirus.

CONTACTS AND LOCATIONS:
Overall Officials: Max W. Sung, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States